CLINICAL TRIAL: NCT06765655
Title: Intraoperative Glucose Monitoring for Diabetes and Stress Hyperglycemia to Reduce Risk of Surgical Site Infections
Brief Title: Perioperative Glucose Monitoring and Treatment to Reduce Risk of Surgical Site Infections and Complications
Acronym: POGM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Peter's Hospital, Albany, NY (Other)
Responsible Party: Principal Investigator, Cheryl Ernst, Cheryl Ernst, MSN, FNP-BC, RNFA, St. Peter's Hospital, Albany, NY
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-1221-4; STUDY00004617 (Other: SUNY Brockport)
Record Dates: First submitted 2025-01-03; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-09

CONDITIONS: Surgical Site Infections; Stress Hyperglycemia
Keywords: Hyperglycemia; Surgical Site infections; Insulin lispro sliding scale; Perioperative monitoring
MeSH Terms: conditions — Surgical Wound Infection; Hyperglycemia | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- POGM (Experimental): Patients will have preoperative Hemoglobin A1C and monitoring of blood glucose every 2 hours during their surgery. If the blood glucose rises over 150 mg/dL, insulin lispro will be administered per sliding scale protocol based on their A1C. Monitoring continues for 48 hours with treatment per protocol as needed.
  Interventions: Drug: Insulin Lispro Injection; Diagnostic Test: glucose testing

INTERVENTIONS:
Drug: Insulin Lispro Injection — point-of-care glucose monitoring via fingerstick perioperatively
  Other Names: POCT glucose testing
Diagnostic Test: glucose testing — POCT glucose testing via fingerstick

SUMMARY:
This study is to determine if glucose monitoring and treatment in surgical procedures over 2 hours help to decrease the surgical site infection risk and reduce postoperative complications. The study uses a preoperative HgBA1C to place patient into a sliding scale insulin category to be used only if the patient has a blood sugar over 150mg/dL during surgery. This is consistent with the CDC recommendation to keep perioperative glucose below 200 mg/dL in surgical patients. The protocol continues for at least 48 hours to treat stress hyperglycemia in non-diabetic patients, and to closely monitor & treat glucose levels in diabetic patients.

DETAILED DESCRIPTION:
Background

Diabetes and variations in glucose control are comorbidities that increase complications in the surgical patient (Harris, 2018). Insulin signaling is impaired during surgery and transient insulin resistance develops. Decreased circulating insulin levels lead to a physiological hyperglycemic response that lasts 24 to 48 hours after surgery. Surgeries involving the chest and abdomen have a longer and more pronounced degree of hyperglycemia reaction in the body (Peacock, 2019). The prevalence of surgical site infections (SSIs) in surgical patients across the United States has gained significant attention as preventable healthcare infections from the Centers for Disease Control and Prevention (CDC) in recent years. A stratified list supporting this evidence was published by the CDC in 1999 titled Prevention of Surgical Site Infection and is the accepted practice guideline for preventing SSIs (Berrios-Torres et al., 2017). The CDC directs surgical specialties to reduce perioperative glycemic control protocol targets to less than 200 mg/dl for all surgical patients to reduce SSIs (Sermkasemskin et al., 2022). Similar evidence-based guidelines were published by the World Health Organization (WHO) and the American College of Surgeons (ACS) (Camperlengo et al., 2023). Nearly six years after these strong guidelines were published, there is still limited evidence that SSI prevention activities are being followed (Camperlengo et al., 2023).

Perioperative stress hyperglycemia is underestimated because of its presumed lower incidence rate compared to diabetes. The rise in patients presenting to surgical facilities with impaired fasting glucose and/or insulin resistance varies from 23 to 60%.

Stress hyperglycemia is summarized as increased glycogenolysis, insulin resistance, and excessive gluconeogenesis in response to neuroendocrine triggers of stress stimulated by the hypothalamic-pituitary-adrenal axis, sympathoadrenal system receptors, and proinflammatory cytokines. The cytokines are tumor necrosis factor-α, interleukin (IL)-1, and IL-6 (Sermkasemsin et al., 2022). Risk factors for stress hyperglycemia include unknown diabetes, a high American Society of Anesthesiologists (ASA) risk score, long surgical duration, blood transfusion, and intraoperative hypotension (Sermkasemskin et al., 2022).

Purpose

The purpose of this DNP project is to focus on reducing postoperative complications by expanding the intraoperative glucose monitoring and treatment protocol to include all surgical patients with procedures lasting over two (2) hours at risk for stress hyperglycemia. The hypothesis is there will be a statistically significant decrease in postoperative complications directly related to longer surgical cases (Peacock, 2019).

Aims and Objectives

Perioperative Glucose Monitoring (POGM) will take place during surgeries that last over two (2) hours St. Peter's Health Partners. The implementation of POGM will occur directly in the operating rooms based on the developed protocol. The review of perioperative data will occur remotely in the outpatient surgical setting through chart reviews by the principal investigator. The objectives of the study are reproducible across all surgical specialties. They include:

1. Obtaining Hemoglobin A1C and blood glucose in enrolled surgical patients preoperatively regardless of diabetes status.
2. Assess blood glucose every two (2) hours perioperatively due to peak action of rapid-release insulin.
3. Institute a standard hyperglycemia treatment protocol via sliding scale rapid acting insulin for any patient with perioperative blood glucose elevations >150 mg/dL.
4. Monitor for postoperative infections, morbidity, and mortality for the sample of enrolled surgical patients for 30 days after surgical intervention. This includes postoperative office visits and phone calls checking on status.

The goal of this study is to lay the groundwork for adapting practice guidelines to meet the modern health needs of our diverse patient population.

Setting

IOGM will occur within the surgical departments of St. Peter's Health Partners (Albany, NY). The implementation of POGM will occur directly in the OR suites based on the developed protocol.

Sample

The pilot study will consist of recruiting adult surgical patients of a participating surgeon. Informed consent is for the collection of patient-related surgical data through medical record review to determine surgical outcomes with POGM. The patient is required to be scheduled for a surgical procedure expected to last 2 hours (120 minutes) at minimum. A power analysis of sample size was made by reviewing random operative cases at SPH in January 2023 through a meta-analysis for this project. The goal is to establish a statistically significant sample size based on probability to avoid a Family-Wise Error Rate that results from incorrect statistical significance related to a sample size that is too large (Thomas & Campbell, 2021). Using a 95% confidence interval and an estimate within 10% of the true proportion of patients that would have intraoperative hyperglycemia, an estimated 76 study participants would be needed.

Target Population

There is currently an inequitable perioperative monitoring of patients based on the Medical Model of Disability. Glucose monitoring perioperatively typically only occurs when there is a known diagnosis of diabetes (DM) per hospital policy. However, the evidence that stress hyperglycemia exists in surgical patients not identified as diabetics contributes to the noted increase in postoperative complications in this population.

Design

The quantitative quasi-experimental research study design yields a high level of descriptive statistical data collected at a ratio/interval level, including the presence of postoperative complications, HgbA1C, and glucose readings. The well-established method of glucose POCT will determine if a patient becomes hyperglycemic during the surgical procedure and can reliably indicate if treatment is needed per hospital protocol. This POCT has strong predictive validity, reflects existing theories, and has strong test/retest reliability (Thomas & Campbell, 2021). From pre-surgery to the end of data collection, the anticipated time to assess the initial impact of the POGM protocol is expected to be approximately 8-12 weeks. This would include initial surgical consultation, an informed consent process, and implementing POGM for each surgical case. Each patient will be monitored for 30 days after surgery for postop complications. The complexity of postop complications is calculated using the Comprehensive Complication Index (CCI) (Hyer et al., 2019)

Data Collection

Quantitative data will be collected during the three (3) perioperative phases via point-of-care (POCT) glucose testing. This monitoring will begin as a pilot test in a select group of surgical patients based on voluntary surgeon enrollment.

Comparison data will be obtained through retrospective analysis of medical records from patients who had surgical procedures >2 hours and occurred before the quality improvement program implementation. A retrospective review of pre- and postoperative POCT glucose levels on the surgical cases of participating surgeons for 2 months prior to implementation of POGM will be performed. Any glucose elevations that may have triggered insulin administration per sliding scale protocol will be noted along with any documented postop SSI occurrence or complication.

ELIGIBILITY:
Inclusion Criteria: Any adult surgical patient who undergoes a procedure expecting to last 2 or more hours regardless of age, gender, race, sex, religion, nation of origin, or other identifiable demographics -

Exclusion Criteria: Type 1 Diabetes or other patients with strick endocrinology orders

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infections | From date of surgery to the end of 30 day postop timeframe
  Assess for the development of superficial, deep, or organ space infections within 30 days of surgery

SECONDARY OUTCOMES:
Postoperative Complications | From date of surgery to the end of 30 day postop timeframe
  Assess for the development and severity of other postoperative complications. Categories include sepsis, cardiac, respiratory, GI, hematologic, Urinary, readmission/reoperation and death.

CONTACTS AND LOCATIONS:
Overall Officials: Jamila Benmoussa, MD, Study Director — St. Peter's Hospital
Locations (1):
- St. Peter's Hospital, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is yet to be determined if the data will be helpful to other researchers